CLINICAL TRIAL: NCT05790577
Title: Comparison of 30% Metformin and 2% Nicotinamide Lotion With Kligman Formula in the Treatment of Melasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ishtiaq Ahmed (Other)
Responsible Party: Sponsor-Investigator, Ishtiaq Ahmed, Ishtiaq Ahmed, Pak Emirates Military Hospital
Organization: Pak Emirates Military Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PakEmiratesMH2
Record Dates: First submitted 2022-08-06; First posted 2023-03-30 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin 30% and 2% Nicotinamispde (Active Comparator): Metformin 30% plus Nicotinamide 2% in the reatment of Melasma
  Interventions: Drug: Metformin and Nicotinamide vs Kligman Formula
- Kligman formula (Active Comparator): Kligman formula in the treatment of Melasma
  Interventions: Drug: Metformin and Nicotinamide vs Kligman Formula

INTERVENTIONS:
Drug: Metformin and Nicotinamide vs Kligman Formula — Comparison of 30% Metformin and 2% Nicotinamide lotion with kligman formula in the treatment of Melasma

SUMMARY:
Comparison of 30% Metformin and 2% Nicotinamide lotion with kligman formula in the treatment of Melasma

DETAILED DESCRIPTION:
A comparative study to evaluate Efficacy and tolerability of new lotion in the treatment of Melasma.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50
* No systemic therapy
* All Co-morbids

Exclusion Criteria:

* Pregnancy
* Age >50
* Taking oral treatment for melasma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Comparison of 30% Metformin and 2% Nicotinamide lotion with kligman formula in the treatment of Melasma | 12 weeks
  Efficacy with measurement of MASI score 4 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Ishtiaq Ahmed, MBBS, Study Director — Pak Emirates Military Hospital
Locations (1):
- PakEmiratesMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No